CLINICAL TRIAL: NCT04376320
Title: Comparison of Two Pre-prosthetic Surgical Techniques for Augmentation of Mandibular Vertical Ridge Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lydia Nabil (Other)
Responsible Party: Sponsor-Investigator, Lydia Nabil, Assistant Professor of Oral and Maxillofacial Surgery, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UAlexandriaDentSurg
Record Dates: First submitted 2020-04-29; First posted 2020-05-06 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Alveolar Ridge Enlargement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1(ceramic membrane) (Active Comparator): using customized ceramic membranes for augmentation of vertical mandibular ridge defects in preparation for implant placement
  Interventions: Device: customised ceramic sheets (Group 1)
- Group 2 (modified sausage technique) (Active Comparator): using tenting titanium screws in conjunction with particulate bone graft and collagen membrane (modified sausage technique) for augmentation of vertical mandibular ridge defects in preparation for implant placement
  Interventions: Combination Product: modified sausage technique (Group 2)

INTERVENTIONS:
Device: customised ceramic sheets (Group 1) — guided bone regeneration
  Arms: Group 1(ceramic membrane)
Combination Product: modified sausage technique (Group 2) — guided bone regeneration
  Arms: Group 2 (modified sausage technique)

SUMMARY:
The aim of this study is to compare two pre-prosthetic surgical techniques for augmentation of vertical mandibular ridge defects in preparation for implant placement, the first using customized ceramic membranes and the second using tenting titanium screws in conjunction with particulate bone graft and collagen membrane (modified sausage technique).

DETAILED DESCRIPTION:
Background: Expansion of the periosteum and soft tissue matrix by tenting has been described as a method of Guided Bone Regeneration (GBR) for reconstruction of atrophic alveolar ridges.

Materials and Methods: The current study is a prospective controlled clinical trial, conducted on 14 patients, having about 7 mm of vertical bone height in the posterior mandible above the inferior alveolar canal. They are divided into 2 equal groups, each consisting of 7 patients. The first group receives customized ceramic membranes with a vertical height 5 mm above the crest of the ridge to tent out the soft tissue matrix, while in the second group, tenting of the soft tissue is done by fixation of two tenting screws, particulate bone graft is packed then covered by collagen membrane that is fixed by bone tacks (modified sausage technique).

ELIGIBILITY:
Inclusion Criteria:

* patients of both genders
* with age range from 40 to 60 years,
* having about 7 mm of vertical bone height in the posterior mandible above the inferior alveolar canal and
* requiring prosthetic rehabilitation with dental implants.

Exclusion Criteria:

* heavy smokers,
* patients undergoing radiotherapy or chemotherapy,
* those having infection or local lesions in the area of surgery, and
* patients with bone diseases which may compromise the results

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-04 (Actual)

PRIMARY OUTCOMES:
mean percentage of change of alveolar bone height | 6 months
  change of alveolar bone height after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No